CLINICAL TRIAL: NCT06623045
Title: Impact of a 12-Week Pelvic Floor Training on Urinary Incontinence in Functional Fitness Training Athletes
Acronym: PFMT-UI-FFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Celia Rodríguez Longobardo, Principal Investigator, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UPM20221125; 20221125 (Other: Universidad Politécnica de Madrid)
Record Dates: First submitted 2024-09-23; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Strength; Muscle Activation; Urinary Incontinence (UI)
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PFM strength (Experimental): This group carries out a 12-week training intervention based on Kegel exercises to improve strength and muscle activation
  Interventions: Other: Pelvic floor muscle training intervention
- Control Group (No Intervention): This group is used as a control group. They keep training their sports discipline but don't join the 12-week PFM training protocol.

INTERVENTIONS:
Other: Pelvic floor muscle training intervention — The training program consisted of 12 weeks of PFM exercises, 3 times per week, with each session lasting between 10 and 15 minutes. The program followed different stages through the weeks: (1) proprioception of pelvic floor muscles activation and integration with diaphragmatic breathing, (2) stabilization and strengthening of the pelvic floor musculature through progressive overloading, and (3) transference of these exercises to FFT practice. During the 12 weeks, short contractions (2") were combined with longer ones (5 to 10"), carrying out the progressive overload by increasing the number of contractions, the duration of the contraction, or by evolving the execution position towards more upright postures and sporting movements.
  Arms: PFM strength

SUMMARY:
Functional fitness training (FFT) is a prominent exercise regimen, that has emerged as the dominant fitness trend of the 21st century , advocating high-intensity exercises with repetitive, impactful movements that often result in increased intra-abdominal pressure (IAP) and neuromuscular fatigue. This demanding training pattern, characterized by minimal rest pauses, has been associated with potential health concerns, particularly urinary incontinence (UI). In athletes, UI is intricately connected to the frequency of exposure to increased IAP during high-impact activities. These activities assume even greater significance in sports, particularly in FFT, where there is an increased frequency of impactful foot contact on the ground and intensive abdominal exercises, potentially correlating with the overload of the pelvic floor muscles and the emergence of dysfunctions. Therefore, this study aims to examine the effects of a 12-week training program focused on Kegel exercises performed with diaphragmatic breathing in nulliparous female FFT athletes. The central hypothesis postulates that after the 12-week intervention, these women will exhibit enhancements in both the muscular activation and contractile capacity of their pelvic floor, leading to a reduction in instances of urine leakage.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous FFT female athletes
* had been practicing FFT or weightlifting for at least 2 years
* train a minimum of 3 days/week
* had not previously performed pelvic floor exercises
* had no medical contraindications or previous pelvic floor surgeries

Exclusion Criteria:

* Any criterion that does not meet the inclusion criteria

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender women
Enrollment: 21 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Strength | From the enrollment to the end of treatment at 12 weeks
  Maximal, medium and minimal force generated of the pelvic floor muscles, measured with a vaginal dynamometer, which involves a pelvimeter probe with two arms that could be separated up to 25°, connected to the Phenix USB2 device (Pelvimètre Phenix, Vivaltis). The closed pelvimeter is inserted into the vagina with one arm positioned against the posterior side of the symphysis pubis. Once in place, to evaluate the contractile force of the PFM, the participant performes a pelvic floor contraction for 10 seconds against the arms of the probe fixed at 5º (an isometric contraction).
muscle activation | From the enrollment to the end of treatment at 12 weeks
  Measured as tone or initial inertia index (III) using a vaginal dynamometer, which involves a pelvimeter probe with two arms that could be separated up to 25°, connected to the Phenix USB2 device (Pelvimètre Phenix, Vivaltis). The closed pelvimeter is inserted into the vagina with one arm positioned against the posterior side of the symphysis pubis. Once in place, the probe is opened by 5° to measure basal muscle activation (initial inertia index) and shock absorption, which assesses the pelvic floor ability to withstand stress.

SECONDARY OUTCOMES:
Urinary incontinence (UI) | From the enrollment to the end of treatment at 12 weeks
  Measured with the International Consultation on Incontinence Questionnaire-short form (ICIQ-SF), which evaluates the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women (in the female athletes in this case). It encompasses 4 items (frequency or urinary incontinence, amount of leakage, overall impact of urinary incontinence and self-diagnostic item) with a scoring scale of 0-21 reflecting the degree of urinary incontinence as slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed anonymously